CLINICAL TRIAL: NCT05154552
Title: Effects of Routine Physical Therapy With and Without Proprioceptive Neuromuscular Facilitation on Balance, Gait and Function in Patients With Parkinson's Disease.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-UOL-FAHS/986/2021
Record Dates: First submitted 2021-11-27; First posted 2021-12-13 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Parkinson Disease
Keywords: Parkinson' disease; Proprioceptive Neuromuscular Facilitation; Freezing of gait; Berg Balance Scale; Functional Independence Measure; Freezing of Gait Questionnaire
MeSH Terms: conditions — Parkinson Disease | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A/ routine physical therapy and PNF (Experimental): In group A, PNF based gait training (15 minutes) and conventional physical therapy (45 minutes) will be performed.
  PNF exercises involved PNF pelvic patterns (pelvic interior elevation and posterior depression), PNF lower extremity D1 Flexion and PNF lower extremity D1 extension (Unilateral during 1st to 3rd week and bilateral from 4th week onwards). Exercises will progress from rhythmic initiation and then progress to slow reversal and agonistic reversal up to 6th week of therapy and continues until 12th week. Each exercise will be repeated for 10 to 20 times.
  Conventional physiotherapy will be administered according to the European Physiotherapy guidelines for Parkinson's disease.
  Other exercises include:
  1. Range of motion exercises
  2. Stretching exercises
  3. Upper and lower limb strengthening exercises
  Interventions: Other: Proprioceptive Neuromuscular Facilitation; Other: Routine physical therapy
- group B/ routine physical therapy (Active Comparator): Conventional physical therapy (45 minute session) will be performed in group B.Conventional physiotherapy will be administered according to the European Physiotherapy guidelines for Parkinson disease.
  Other exercises include:
  1. Range of motion exercises
  2. Stretching exercises
  3. Upper and lower limb strengthening exercises
  Interventions: Other: Routine physical therapy

INTERVENTIONS:
Other: Proprioceptive Neuromuscular Facilitation — Proprioceptive Neuromuscular Facilitation (PNF) is a more advanced form of flexibility training, which involves both the stretching and contracting of the muscle group being targeted. PNF stretching is one of the most effective forms of stretching for improving flexibility and increasing range of motion.
  Arms: group A/ routine physical therapy and PNF
Other: Routine physical therapy — Routine physiotherapy in Parkinson Disease will be administered according to the European Physiotherapy guidelines for Parkinson Disease and focused on the following areas based on the stage of the disease:Self-management support, prevention of inactivity and fear of falls, maintaining or improving global motor activities, improvement of physical performance, and improvement in the ability to perform transfer, balance, gait, and manual activities, reduce pain, and delay the onset of physical limitations.
  Other exercises include:
  1. Range of motion exercises
  2. Stretching exercises
  3. Upper and lower limb strengthening exercises

SUMMARY:
Objective of this study is to compare the effectiveness of routine physical therapy with and without Proprioceptive Neuromuscular Facilitation on Balance, gait and function in patients with Parkinson's disease.

Alternate hypothesis:

There will be a difference in the effects of routine physical therapy with and without proprioceptive neuromuscular facilitation on balance, gait and function in patients with Parkinson's disease.

Null hypothesis:

There will be no difference in the effects of routine physical therapy with and without proprioceptive neuromuscular facilitation on balance, gait and function in patients with Parkinson's disease.

DETAILED DESCRIPTION:
It will be a prospectively registered, parallel designed, single blinded randomized controlled trial with concealed allocation, conducted in University of Lahore Teaching Hospital and Sir Ganga Raam hospital, Lahore, Pakistan. Patients who met eligibility criteria will be informed about the aim of study.consent form will be signed by all eligible participants. Eligibility of participants will be confirmed by the physiotherapist of research team before randomization. After baseline assessment, eligible patients will be randomly allocated(in a 1:! ratio) in two groups( group A and group B). Fish bowl method of randomization will be used and will be done by one of the research team members who will not involve in patient recruitment or assessment or data analysis.

Randomization assignments will be kept in opaque, sealed envelopes for concealment of group allocation and will be unsealed by researcher after baseline testing. Researchers who assess outcomes or will do data analyses will be masked to group allocation.The calculated sample size is 32 (16 in each group), after adding 20% dropout the sample size will be 32+6=38, 19 patients in each group.(statistical power 80% and alpha level of 5%).

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients of age between 60 and 85 years, diagnosed with Parkinson's disease by a neurologist.
* Patients with Hoehn and Yahr stages 1-3.
* Patients with a stable drug program and acclimated to their current medication use for at least 2 weeks.

Exclusion Criteria:

* Cognitive deficits (scores of <26 on the Mini-Mental State Examination).
* Moderate or severe depression (scores of >17 on the Beck Depression Inventory).
* Patients with neurological diseases, arthrosis, or total hip joint replacement.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2022-03-03 (Actual)

PRIMARY OUTCOMES:
Berg balance scale (BBS) (to access the change in ability to balance in individuals at baseline, 6th and 12th week of interventions.) | the change in ability to balance in individuals at baseline, 6th and 12th week of interventions.
  It is used to objectively determine a patient's ability or inability to safely balance during a series of predetermined tasks. It consist of a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4.0 denotes inability to complete the item, and 4 the ability to accomplish the task. Scores of less than 45 out of 56 are accepted as indicative of balance disorders in the elderly.
The Freezing of Gait Questionnaire (FOGQ) (to access the change in freezing of gait in individuals at baseline, 6th and 12th week.) | the change in freezing of gait in individuals at baseline, 6th and 12th week
  It is used to assess freezing of gait severity in patients with Parkinson's disease. It consists of a 6-item questionnaire. A 5-point scale is used to mark scores. Zero (absence of symptoms) to 4 (most severe), is used for each item to rank severity of symptoms.
Functional Independence Measure (FIM) (to assess the change in ability to do activities of daily living at baseline, 6th and 12th week.) | the change in ability to do activities of daily living at baseline, 6th and 12th week
  It is used to assess the ability of patients to do activities of daily living. It consist of 18-item, clinician-reported scale that assesses function in six areas including self-care, continence, mobility, transfers, communication, and cognition. Total score for FIM will be a value between 18 and 126. Higher the score, more independent the patient is.

CONTACTS AND LOCATIONS:
Overall Officials: Tahzeeb Mazhar, MSPTN, Principal Investigator — University of Lahore, Pakistan
Locations (2):
- Pakistan (2):
  - Sir Ganga Raam Hospital, Lahore, Punjab Province
  - University of Lahore Teaching Hospital, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: Undecided